CLINICAL TRIAL: NCT05096104
Title: Patient Satisfaction During Artificial Induction of Labor by Cervical Ripening
Acronym: CERVICAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8294
Record Dates: First submitted 2021-08-06; First posted 2021-10-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cervical Ripening
Keywords: Cervical Ripening; PREGNANCY; LABOR INDUCED; Artificial induction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
20% of deliveries take place following an artificial induction of labor. The latter sometimes requires prior cervical ripening, of which the two most widely used methods in France are oral misoprostol and the balloon catheter, left to the discretion of clinicians.

The objective of this study is to observe which cervical maturation method patients choose when an artificial induction of labor with an unfavorable cervical status must be carried out, and to observe the patient's criteria as to the choice made, as well as their experience and their satisfaction with artificial induction of labor, in order to improve our clinical practices, the experience of childbirth, and promote patient autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years old)
* Patient who underwent induction of labor between February 1, 2020 and February 29, 2021
* Patient not having expressed her opposition, after information, to the reuse of her data for the purposes of this research.

Exclusion Criteria:

* Patient who expressed her opposition to participating in the study
* Absence of prior cervical maturation (Bishop score greater than or equal to 6 on the day of initiation)
* Gestational age less than 37 weeks, multiple pregnancy, scarred uterus, non-cephalic presentation, death in utero and severe fetal malformation (requiring neonatal resuscitation or with a palliative care plan)
* Patient for whom the triggering method was chosen by the practitioner
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman who underwent induction of labor between February 1, 2020 and February 29, 2021
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the cervical ripening method that patients choose when artificial induction of labor with unfavorable cervical status must be performed | Files analysed retrospectively from JFebruary 01, 2020 to February 29, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas SANANES, MD, PhD, Principal Investigator — Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France